CLINICAL TRIAL: NCT02025218
Title: Iressa Re-challenge in Advanced NSCLC EGFR Mutated Patients Who Responded to an EGFR-TKI Used as First-line or Previous Treatment (NVALT 16)
Brief Title: Iressa Re-challenge in Advanced NSCLC EGFR-mutated Patients
Acronym: IRENE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Justine Kuiper, MD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRENE study - NVALT 16
Record Dates: First submitted 2013-12-23; First posted 2013-12-31 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: NSCLC; EGFR; TKI; Re-challenge; Lung Cancer; Resistance
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Re-administration gefitinib (Experimental)
  Interventions: Drug: Gefitinib standard dose

INTERVENTIONS:
Drug: Gefitinib standard dose

SUMMARY:
To evaluate the effect of re-administration of gefitinib to EGFR-mutated NSCLC patients who had been treated with at least one line of TKIs followed by another line of treatment (non-TKI)

DETAILED DESCRIPTION:
Rationale: Gefitinib is a registered first-line treatment for EGFR-mutated NSCLC patients. There is a lack of evidence for second and third line therapies in this category of patients. Several case reports have described successful re-administration of gefitinib to NSCLC patients who achieved objective response with the initial administration of gefitinib before eventual progression.

Objective: The primary objective of this study is to evaluate the disease control rate (DCR; confirmed complete response (CR) or partial response (PR), or stable disease (SD)) of gefitinib using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 in patients with activating sensitising Epidermal Growth Factor mutation positive (EGFR M+) NSCLC. The secondary objectives of the study are: objective response rate (ORR) according to RECIST, progression free survival (PFS) according to RECIST, overall Survival (OS), EGFR Mutational status of tumour tissue both activating and resistance EGFR mutations analysis and the association between the Veristrat assay (Biodesix) and both PFS and OS will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC with an activating sensitising EGFR TK mutation as determined before starting the first EGFR-TKI treatment by using a well-validated and robust methodology
* Female or male patients aged 18 years or over with locally advanced or metastatic stage IIIB/IV disease, not suitable for therapy of curative intent or stage IV (metastatic) disease, eligible for gefitinib re-challenge treatment for NSCLC who have already received an EGFR-TKI with a documented complete (CR) or partial response (PR) or stable disease (SD) >12 weeks as the best response to their 1st EGFR-TKI treatment and who have received any subsequent anti-cancer therapy (excluding EGFR-TKIs) treatment, including but not limited to doublet platinum based chemotherapy or docetaxel monotherapy or pemetrexed monotherapy, on which they progressed.
* Measurable disease defined as at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with spiral CT or MRI and which is suitable for accurate repeated measurements.
* WHO / ECOG / Zubrod performance status 0-2.
* Possibility of obtaining tumour material before the start of the study treatment.

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of the product treatment with no persistent radiation toxicity. Previous adjuvant chemotherapy is allowed.
* Progressive disease or stable disease (SD) <12 weeks as best response to the 1st line treatment with an EGFR-TKI
* Consideration to require radiotherapy to the lung at the time of study entry or in the near future
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease. Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline
* Known or suspected brain metastases or spinal cord compression, unless treated with surgery and/or radiation.
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Concomitant use of known CYP 3A4 inducers such as phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort
* Pregnancy or breast-feeding
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (eg, unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Other co-existing malignancies or malignancies diagnosed within the last 2 years with the exception of basal cell carcinoma or cervical cancer in situ
* Life expectancy of less than 12 weeks
* Treatment with a non-approved or investigational drug within 30 days before day 1 of study treatment
* Involvement in the planning and/or conduct of the study (applies to both NVALT staff or staff at the study site)
* Previous enrolment or treatment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Disease control rate | 6 months after last included patient

CONTACTS AND LOCATIONS:
Locations (14):
- Netherlands (14):
  - Ziekenhuis Groep Twente, Almelo
  - VU University medical Center, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Wilhelmina Ziekenhuis Assen, Assen
  - Rode Kruis ziekenhuis, Beverwijk
  - Deventer ziekenhuis, Deventer
  - Gelderse vallei, Ede
  - Catharina ziekenhuis, Eindhoven
  - Martini ziekenhuis, Groningen
  - University Medical Center Groningen, Groningen
  - Canisius Wilhelmina ziekenhuis, Nijmegen
  - Maasstad ziekenhuis, Rotterdam
  - VieCurie Hospital, Venlo
  - Isala klinieken, Zwolle